CLINICAL TRIAL: NCT00258518
Title: Estimation of Respiratory Mechanics (Respiratory System, Chest Wall and Lung Elastance) and Pleural Effusion at the Bedside With CT Scan.
Brief Title: Respiratory Mechanics and Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 1500
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Critically Ill; Acute Lung Injury; ARDS
Keywords: Critically ill patients
MeSH Terms: conditions — Critical Illness; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: ALI/ARDS patients
  Interventions: Procedure: mechanical ventilation/CT Scan

INTERVENTIONS:
Procedure: mechanical ventilation/CT Scan — evaluation of pleural effusion and respiratory mechanics, CT scan

SUMMARY:
The investigators aim to compare the respiratory mechanics in acute lung injury (ALI)/acute respiratory diseases syndrome (ARDS) patients with and without pleural effusion.

DETAILED DESCRIPTION:
In ALI/ARDS we evaluated the respiratory mechanics (respiratory system, chest wall and lung elastance) at the bedside while pleural effusion was evaluated with CT scan. Thus we will be able to estimate any possible role of pleural effusion on the respiratory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* ALI/ARDS patients underwent invasive mechanical ventilation

Exclusion Criteria:

* Haemodynamic instability
* Chronic obstructive pulmonary disease (COPD) patients

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALI/ARDS patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Role of pleural effusion and respiratory mechanics | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy